CLINICAL TRIAL: NCT02911389
Title: Unsupervised Home Exercise With and Without a Web-based Recovery Platform as Compared to Traditional Outpatient Physiotherapy After Total Knee Arthroplasty: A Prospective, Randomized Controlled Trial
Brief Title: Home PT vs FORCE PT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 16Chen01
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (3):
- Home PT via web-based platform (Active Comparator): unsupervised, home rehabilitation delivered by a web-based platform
  Interventions: Other: Home PT via web-based platform
- Home PT via paper manual (Active Comparator): unsupervised, home rehabilitation delivered by a paper manual
  Interventions: Other: Home PT via paper manual
- outpatient PT (Active Comparator): outpatient physical therapy
  Interventions: Other: outpatient PT

INTERVENTIONS:
Other: Home PT via web-based platform
  Arms: Home PT via web-based platform
Other: Home PT via paper manual
  Arms: Home PT via paper manual
Other: outpatient PT
  Arms: outpatient PT

SUMMARY:
The purpose of this study is to determine if unsupervised, home rehabilitation delivered by a web-based platform or paper manual is a safe and effective alternative to outpatient physical therapy after total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient undergoing unilateral, primary TKA

Exclusion Criteria:

1. Patients without access to the Internet
2. Patients without access to outpatient PT
3. Revision or conversion TKA
4. Patients discharged to a rehabilitation unit or other form of respite care such as a skilled nursing facility, acute rehabilitation center, convalescent home, long-term care facility or nursing home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Knee Range of Motion | 1 month post surgery
  Measured in degrees from 0-130

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States